CLINICAL TRIAL: NCT03337217
Title: Colonoscopy in the Prone Position for Patients With BMI Greater Than 30 Is Superior to Standard Left Lateral Decubitus Position
Brief Title: Colonoscopy in the Prone Position for Patients With BMI Greater Than 30
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Brooke Corning, Principal Investigator, Fellow Physician, Dept of Internal Medicine Division of Gastroenterology and Hepatology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20078
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Obesity
Keywords: colonoscopy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Position (Experimental): Position during colonoscopy
  Interventions: Procedure: Position during colonoscopy
- Left lateral decubitus position (Active Comparator): Position during colonoscopy
  Interventions: Procedure: Position during colonoscopy

INTERVENTIONS:
Procedure: Position during colonoscopy — Position during colonoscopy

SUMMARY:
In the United States, colonoscopy has become the most commonly used screening test for colorectal cancer. Colonoscopy is typically performed with the patient starting in the left lateral decubitus position, however there is little data to support this practice and starting position is variable amongst individual gastroenterology physicians.

The investigators plan to randomize patients with Body Mass Index >30 that are presenting to the University of Virginia for colonoscopy to either the prone or left lateral decubitus position. The investigators will then record and compare cecal intubation times as well as amount of sedation used and complications to help determine which position is superior for this patient population.

DETAILED DESCRIPTION:
Patients that have been scheduled for colonoscopy will undergo chart review. Patients who meet inclusion criteria will be invited to participate at the time consent is obtained for the colonoscopy. Participants will then be randomized to one of two colonoscopy starting positions.

After randomization, patients will begin the colonoscopy in either the prone position or left lateral decubitus position.

It is common practice to re-position the patient during endoscopy (including supine and prone positions) and some endoscopists commonly employ prone starting position for obese patients, although there is no estimate in the literature as to the prevalence of this practice.

No additional interventions will be performed for research purposes. During the colonoscopy, the endoscopist will be allowed, as usual, to adjust patient position as needed to complete the procedure. Cecal intubation time, amount of sedation used, and any intra-procedural complications (hypoxia, hypotension, etc) will be recorded for data analysis. This information is standardly recorded in the procedure report in the patient's medical record. The study will not affect any interventions performed during the colonoscopy such as polyp removal or biopsies as, clinically indicated. Per endoscopy unit protocol, patients will be monitored in the recovery area and discharged home with supervision. The study requires no further direct patient interaction after the colonoscopy is completed. Charts will be reviewed at 30 days to assess for any delayed and unexpected complications.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30
* Undergoing screening or diagnostic colonoscopy with conscious sedation

Exclusion Criteria:

* Pregnant women (self reported).
* Cognitively impaired patients
* History of colonic resection
* Cannot lay in prone position
* History of colon malignancy
* Procedure aborted due to inadequate bowel prep
* Severe pulmonary problems (including baseline oxygen use)
* Inability to provide consent for themselves

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Cecal intubation time measured in seconds | Measured once during colonoscopy.
  Time to advance the colonoscope to the cecum during colonoscopy.

SECONDARY OUTCOMES:
Milligrams of sedative used for sedation | Measured once at the completion of the colonoscopy.
  Amount of fentanyl and midazolam needed for adequate sedation.
Technical difficulty of procedure (questionnaire) | Recorded once at the completion of the colonoscopy.
  Measure of subjective sense of difficulty as perceived by the endoscopist.

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Corning, MD, Principal Investigator — University of Virginia, Dept of Internal Medicine, Divison of Gastroenterology and Hepatology
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uddin FS, Iqbal R, Harford WV, Dunbar KB, Cryer BL, Spechler SJ, Feagins LA. Prone positioning of obese patients for colonoscopy results in shortened cecal intubation times: a randomized trial. Dig Dis Sci. 2013 Mar;58(3):782-7. doi: 10.1007/s10620-012-2468-x. Epub 2012 Nov 10. PMID 23143737
- [Background] Weinstock LB, Early DS. Colonoscopy in the tilt-down position. Gastrointest Endosc. 2014 Oct;80(4):746. doi: 10.1016/j.gie.2014.05.328. No abstract available. PMID 25220519
- [Background] Rex DK. Achieving cecal intubation in the very difficult colon. Gastrointest Endosc. 2008 May;67(6):938-44. doi: 10.1016/j.gie.2007.12.028. No abstract available. PMID 18440383
- [Background] De Silva AP, Kumarasena RS, Perera Keragala SD, Kalubowila U, Niriella M, Dassanayake AS, Pathmeswaran A, de Silva HJ. The prone 12 o'clock position reduces ileal intubation time during colonoscopy compared to the left lateral 6 o'clock (standard) position. BMC Gastroenterol. 2011 Aug 4;11:89. doi: 10.1186/1471-230X-11-89. PMID 21816067
- [Background] Vergis N, McGrath AK, Stoddart CH, Hoare JM. Right Or Left in COLonoscopy (ROLCOL)? A Randomized Controlled Trial of Right- versus Left-Sided Starting Position in Colonoscopy. Am J Gastroenterol. 2015 Nov;110(11):1576-81. doi: 10.1038/ajg.2015.298. Epub 2015 Sep 29. PMID 26416195
- [Background] Lucendo AJ. Colonoscopy in obese patients: time to change position. Dig Dis Sci. 2013 Mar;58(3):608-9. doi: 10.1007/s10620-012-2542-4. Epub 2013 Jan 12. No abstract available. PMID 23314857
- [Background] Lieberman DA, Rex DK, Winawer SJ, Giardiello FM, Johnson DA, Levin TR. Guidelines for colonoscopy surveillance after screening and polypectomy: a consensus update by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2012 Sep;143(3):844-857. doi: 10.1053/j.gastro.2012.06.001. Epub 2012 Jul 3. No abstract available. PMID 22763141
- [Background] Flegal KM, Kruszon-Moran D, Carroll MD, Fryar CD, Ogden CL. Trends in Obesity Among Adults in the United States, 2005 to 2014. JAMA. 2016 Jun 7;315(21):2284-91. doi: 10.1001/jama.2016.6458. PMID 27272580
- [Background] Witte TN, Enns R. The difficult colonoscopy. Can J Gastroenterol. 2007 Aug;21(8):487-90. doi: 10.1155/2007/520431. No abstract available. PMID 17703247

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT03337217/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT03337217/ICF_001.pdf